CLINICAL TRIAL: NCT02332382
Title: The Influence of Mother Nutrition on the Composition of Fatty Acid, Oligosacharides and Its Effect on Breast Milk Microbiome
Brief Title: The Influence of Mother Nutrition on Breast Milk Microbiome
Acronym: Breast Milk
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Yoram Bujanover MD, Head pediatric gastroenterology service, Sheba Medical Center
Other Study IDs: 1424-14-SMC
Record Dates: First submitted 2015-01-04; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Breast Milk, Composition, Microbiome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months

SUMMARY:
The research subject

Health organizations around the world have determined that breastfeeding is the most critical source of nutrition for newborns in the first weeks and months of their lives. A mother's breast milk contains unique nutritious components and other nonnutritive elements that help promote healthy baby growth and development (1, 2). Recent studies show that a mother's breast milk contains components that vary from each specimen. There are great evidences that maternal and environmental factors have a strong influence on the composition of breast milk. Fatty acids, the second most common component found in breast milk, show extreme sensitivity to maternal nutrition (3, 4).

Latest studies show that breast milk also contains bacterial communities that may have health implications of newborn. The structure of these bacterial communities also varied greatly between subjects (5) .

In the research, we propose to investigate the connection between maternal nutrition, different fatty acids and their role in the growth and development of bacterial populations existing in breast milk.

ELIGIBILITY:
Inclusion Criteria:Healthy lactating women, breast feeding for the first 3 months after delivery

Exclusion Criteria: No compliance, sickness, drug consumption

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy lactating women
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Change in breast milk composition in relation to nutritional intake | 3 months